CLINICAL TRIAL: NCT05405842
Title: Effects of Transauricular Vagal Nerve Stimulation on Electrogastrography (EGG) and Heart Rate Variability (HRV) in Healthy Subjects, Functional Dyspepsia, and Gastroparesis
Brief Title: Transauricular Vagal Nerve Stimulation; Functional Dyspepsia and Gastroparesis
Acronym: AVNS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There were equipment issues with the vendor that could not be resolved; therefore, enrollment was never opened.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Linda Nguyen, Clinical Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63421
Record Dates: First submitted 2022-05-23; First posted 2022-06-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gastroparesis; Functional Dyspepsia; Healthy; Digestive System Disease; Gastroenterology
Keywords: vagal nerve stimulation; EGG; gastroparesis; functional dyspepsia; auricular; stanford; digestive; gastroenterology
MeSH Terms: conditions — Gastroparesis; Digestive System Diseases | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: n= 60 3 groups : gastroparesis (n=20); functional dyspepsia (n=20) ; health controls (n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Gastroparesis (Experimental): Patients diagnosed with Gastroparesis.
  Interventions: Device: Transauricular Vagal Nerve Stimulation
- Functional Dsypepsia (Experimental): Patients diagnosed with Functional Dsypepsia.
  Interventions: Device: Transauricular Vagal Nerve Stimulation
- Healthy Controls (Experimental): Healthy volunteers (without Functional Dsypepsia or Gastroparesis)
  Interventions: Device: Transauricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transauricular Vagal Nerve Stimulation — TENS 7000 is a handheld device used to deliver electrical impulses for nerve stimulation to help modulate and treat chronic pain. The manufacturer, Roscoe, has regulatory approval for the use of nerve stimulator therapy in the acute and/or prophylactic treatment of headaches, migraines, sciatica, muscle spasms, acute and chronic pain, and improve circulation. It is FDA approved in the USA for the above indications, but has not been approved for use in gastrointestinal diseases such as gastroparesis or functional dyspepsia. It has been registered as an investigational new device in various clinical trials. The purpose of this protocol is to provide vagal nerve stimulation to patients with gastroparesis, functional dyspepsia, and healthy controls as a comparison.
  Other Names: vagal nerve stimulation

SUMMARY:
The goal of this study is to establish parameters of gastric myoelectrical activity and heart rate variability in healthy human subjects and compare and contrast them to those with gastroparesis and functional dyspepsia, at baseline and following taVNS.

DETAILED DESCRIPTION:
This is a prospective pilot study assessing the relationship of electrogastrography and heart rate variability, with transauricular stimulation of the vagal nerve in healthy subjects compared to gastroparesis and functional dyspepsia patients. The investigators plan to recruit a total of 60 patients: 20 healthy volunteers, 20 gastroparesis, and 20 functional dyspepsia patients. Participants will undergo two testing sessions in which electrogastrography (EGG) and heart rate variability (HRV) will be measured using electrodes following transauricular vagal nerve stimulation (tAVNS) at various frequencies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age 18-85 years.
3. Healthy volunteer or established diagnosis of idiopathic, diabetic, or postsurgical gastroparesis and functional dyspepsia.
4. Patient is capable of giving informed consent.
5. Patient is on stable doses of other medications for gastroparesis or functional dyspepsia for preceding 4 weeks prior to enrollment (including cholinergics, anti-cholinergics, dopamine and serotonin receptor agonists/antagonists, motility agents, neuromodulators, herbals).

Exclusion Criteria:

1. Any diagnosis of systemic autonomic dysfunction.
2. Use of narcotic, anticholinergic, cholinergic, or promotility medications in preceding 2 weeks of study.
3. Enteric feeding tubes.
4. Parenteral nutrition.
5. Severe disease flare requiring hospitalization or ER visits within 3 months of study.
6. Untreated depression or suicidal thoughts.
7. Pregnant/breastfeeding women.
8. History of gastric pacemaker implantation.
9. Implantable electronic devices (i.e. cardiac pacemakers)
10. Extrinsic myopathy/neuropathy
11. Vagal nerve injury.
12. High risk cardiac arrhythmias (high grade AV block, atrial fibrillation, atrial flutter).
13. GERD.
14. History of dumping syndrome.
15. History of rapid gastric emptying.
16. Severe allergy to skin adhesives.
17. Concurrent enrollment in other clinical trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Establish EGG/HRV parameters and effects following taVNS | 3-5 years
  The first primary outcome measure will be to establish measures of EGG and HRV parameters in healthy volunteers and determine effects of tAVNS on EGG and HRV. The HRV parameters to be measured will include mean heart rate (HR), standard deviation of HR, mean respiratory rate (RR) interval, standard deviation of RR interval, low/high frequency (LF, HF, LF/HF), normalized LF, and normalized HF. The EGG parameters to be measured will be of gastric slow wave power, gastric slow wave propagation, and phase gradient directionality.

SECONDARY OUTCOMES:
Determine deviations in EGG/HRV parameters and effects following taVNS | 3-5 years
  To determine if gastroparesis or functional dyspepsia patients have significant deviations in EGG (slow wave power, propagation, and phase gradient directionality) and HRV (mean HR, LF, HF, mean RR) parameters at baseline and following tAVNS compared to healthy volunteers.

OTHER OUTCOMES:
Determine Stimulation Parameters of tAVNS with Greater Effect on Gastroparesis and Functional Dyspepsia | 3-5 years
  To determine what stimulation parameters have a greater effect on EGG variables (gastric slow wave power, propagation, and phase gradient directionality,) and HRV variables (mean HR, mean RR, LF, HF) in gastroparesis and functional dyspepsia patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy XY Zhou, DO, Study Director — Fellow; Sandya Subramanian, Phd, Principal Investigator — Postdoctoral Fellow; Todd Coleman, Phd, Principal Investigator — Associate Professor; Linda Nguyen, MD, Principal Investigator — Clinical Professor of Medicine

IPD SHARING:
Plan to Share IPD: No